CLINICAL TRIAL: NCT07351227
Title: Comparison of the Effectiveness and Cost-Effectiveness of McGRATH™ MAC and Besdata Videolaryngoscopes in the Orotracheal Intubation of Children: A Non-Inferiority Randomized Clinical Trial
Brief Title: Pediatric Airway: Noninferiority Trial of Devices for Intubation Assessment
Acronym: PANDA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Vinícius C Quintão, MD, MSc, PhD, Assistant Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: PANDA
Record Dates: First submitted 2026-01-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Intubation, Intratracheal; Airway Management; Video Laryngoscope; Cost Effectiveness
Keywords: Videolaryngoscope; Pediatric orotracheal intubation; Cost effectiveness; McGrath MAC; BESDATA
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blind clinical trial designed to evaluate the cost-effectiveness and clinical outcomes of the BESDATA BD-DF and McGrath™ MAC videolaryngoscopes in pediatric patients under one year of age undergoing elective surgery under general anesthesia requiring orotracheal intubation.
  Inclusion criteria The study will include children aged between 6 months and 3 years who are scheduled for elective surgery under general anesthesia at the Children's Institute (Instituto da Criança - ICr) of the Hospital das Clínicas Complex, University of São Paulo Medical School (HC-FMUSP), provided that informed consent is obtained from their parents or legal guardians.
  Exclusion criteria Patients under one year of age will be excluded if informed consent is not obtained from their legal guardians, if they are classified as ASA physical status IV or higher, present with hemodynamic instability, or have craniofacial abnormalities or oral deformities suggestive of a po
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- McGrath MAC (Active Comparator): Intubation the included participants with the McGrath MAC videolaryngoscope
  Interventions: Device: Intubation
- BESDATA BD-DF (Experimental): Intubation the included participants with the BESDATA BD-DF videolaryngoscope
  Interventions: Device: Intubation

INTERVENTIONS:
Device: Intubation — Intubation of pediatric patients under one year of age undergoing elective surgery under general anesthesia requiring orotracheal intubation, with one or another videolaryngoscope device.

SUMMARY:
The goal of this clinical trial is to find out whether the BESDATA BD-DF videolaryngoscope works as well as the McGRATH™ MAC videolaryngoscope for placing a breathing tube in infants during surgery. The study will also compare the costs associated with using each device.

The main questions this study aims to answer are:

Is the BESDATA BD-DF videolaryngoscope as effective as the McGRATH™ MAC videolaryngoscope for successful placement of a breathing tube on the first attempt in infants?

Are there differences between the two devices in terms of procedure time, number of attempts, airway-related complications, and overall costs?

Researchers will compare infants who are intubated using the BESDATA BD-DF videolaryngoscope with infants who are intubated using the McGRATH™ MAC videolaryngoscope to see whether the two devices perform similarly and whether one is more cost-effective than the other.

Participants will:

Be randomly assigned to have a breathing tube placed using one of the two videolaryngoscopes;

Receive standard general anesthesia for an elective surgical procedure;

Have information collected during and after the procedure to assess safety, effectiveness, and costs.

DETAILED DESCRIPTION:
Airway management in infants and young children is technically challenging and carries a higher risk of complications than in older pediatric or adult patients. Achieving successful orotracheal intubation on the first attempt is particularly important in this population due to limited oxygen reserves and increased vulnerability to hypoxia, airway trauma, and hemodynamic instability. Videolaryngoscopy has been introduced as an alternative to conventional direct laryngoscopy with the potential to improve glottic visualization and intubation success. However, evidence comparing different videolaryngoscopy devices in infants remains limited, and there is currently no consensus regarding the optimal device for this age group.

Although several videolaryngoscopes are available on the market, most comparative studies have focused on adult populations. In pediatrics, and especially in infants under one year of age, published data are scarce. The McGRATH™ MAC videolaryngoscope has been more extensively studied and is widely used in clinical practice. In contrast, the BESDATA BD-DF videolaryngoscope is a newer device with very limited clinical evidence, and no head-to-head trials have compared it with other videolaryngoscopes in children. Furthermore, despite the increasing adoption of videolaryngoscopy, the economic impact of using different devices has not been adequately investigated in pediatric settings.

This study is designed to address these gaps by comparing the clinical performance and cost-effectiveness of the BESDATA BD-DF and McGRATH™ MAC videolaryngoscopes in infants undergoing elective surgery under general anesthesia. The trial will evaluate whether the BESDATA device is non-inferior to the McGRATH device in terms of intubation effectiveness while also assessing relevant economic outcomes associated with each technology.

The study will be conducted as a prospective, randomized, double-blind clinical trial at a tertiary pediatric center. Participants will be randomly allocated to undergo tracheal intubation with one of the two videolaryngoscopes. All procedures will be performed by trained anesthesiologists experienced with both devices, and data will be collected using a standardized protocol in a secure electronic database.

In addition to comparing clinical performance, the study will include an economic evaluation that considers the costs of device acquisition, required consumables, and expenses related to potential postoperative complications associated with airway management. This integrated approach aims to provide clinically meaningful and economically relevant information to support evidence-based decision-making in pediatric anesthesia.

By directly comparing two videolaryngoscopy systems in a randomized design, this trial seeks to generate high-quality evidence regarding the most effective and sustainable option for airway management in infants. The results are expected to inform clinical practice, guide resource allocation, and contribute to safer perioperative care for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* The study will include children aged between 6 months and 3 years who are scheduled for elective surgery under general anesthesia at the Children's Institute (Instituto da Criança - ICr) of the Hospital das Clínicas Complex, University of São Paulo Medical School (HC-FMUSP), provided that informed consent is obtained from their parents or legal guardians.

Exclusion Criteria:

* Patients under one year of age will be excluded if informed consent is not obtained from their legal guardians, if they are classified as ASA physical status IV or higher, present with hemodynamic instability, or have craniofacial abnormalities or oral deformities suggestive of a potentially difficult airway.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 226 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
First-attempt intubation success | From randomization until up to 15 minutes
  Proportion of participants in whom successful orotracheal intubation is achieved on the first laryngoscopy attempt using the allocated videolaryngoscope, without the need for additional attempts or device change.

SECONDARY OUTCOMES:
Incremental cost-effectiveness ratio of videolaryngoscopes | From the day of surgery until hospital discharge (up to 30 days postoperatively)
  Cost-effectiveness will be assessed using the Incremental Cost-Effectiveness Ratio (ICER), calculated as the difference in total cost per patient (unit: US dollars) between the BESDATA BD-DF and McGRATH™ MAC devices divided by the difference in effectiveness, defined as the rate of successful first-attempt intubation (unit: percentage). Total costs will include device and consumable expenses and direct hospital costs related to postoperative complications and additional length of stay.

OTHER OUTCOMES:
Number of intubation attempts | During anesthetic induction
  Number of intubation attempts
Cormack-Lehane grade | During anesthetic induction
  Cormack-Lehane grade
Percentage of glottic opening (POGO) score | During anesthetic induction
  Percentage of glottic opening (POGO) score
Intubation-related complications. | During anesthetic induction
  Intubation-related complications, including mechanical trauma and desaturation;

CONTACTS AND LOCATIONS:
Overall Officials: Vinícius C Quintão, MD, PhD, Principal Investigator — Hospital das Clínicas HCFMUSP
Locations (1):
- Instituto da Criança e do Adolescente, Hospital das Clinicas HCFMUSP, Faculdade de Medicina, Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No, individual participant data will not be shared.

REFERENCES:
- [Background] Gupta A, Sharma R, Gupta N. Evolution of videolaryngoscopy in pediatric population. J Anaesthesiol Clin Pharmacol. 2021 Jan-Mar;37(1):14-27. doi: 10.4103/joacp.JOACP_7_19. Epub 2021 Apr 10. PMID 34103817
- [Background] Fiadjoe JE, Nishisaki A, Jagannathan N, Hunyady AI, Greenberg RS, Reynolds PI, Matuszczak ME, Rehman MA, Polaner DM, Szmuk P, Nadkarni VM, McGowan FX Jr, Litman RS, Kovatsis PG. Airway management complications in children with difficult tracheal intubation from the Pediatric Difficult Intubation (PeDI) registry: a prospective cohort analysis. Lancet Respir Med. 2016 Jan;4(1):37-48. doi: 10.1016/S2213-2600(15)00508-1. Epub 2015 Dec 17. PMID 26705976
- [Background] Hu X, Jin Y, Li J, Xin J, Yang Z. Efficacy and safety of videolaryngoscopy versus direct laryngoscopy in paediatric intubation: A meta-analysis of 27 randomized controlled trials. J Clin Anesth. 2020 Nov;66:109968. doi: 10.1016/j.jclinane.2020.109968. Epub 2020 Jul 6. PMID 32645564
- [Background] Abbas A, Samad L. Children at the heart of global surgery: children's surgery in low- and middle-income countries. J Public Health Emerg 2020;4:34.10.21037/jphe-2020-gs-08
- [Background] Rabbitts JA, Groenewald CB. Epidemiology of Pediatric Surgery in the United States. Paediatr Anaesth. 2020 Oct;30(10):1083-1090. doi: 10.1111/pan.13993. Epub 2020 Aug 29. PMID 32777147